CLINICAL TRIAL: NCT04541147
Title: A Randomized Control Trial of Post-operative Course of Oral Dexamethasone and Effect on Opioid Usage in Pediatric Tonsillectomies in a Tertiary Care Center
Brief Title: Opioid & Steroid Use Following Tonsillectomy in Pediatric Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00103025
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone; Analgesics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dexamethasone plus analgesics (Experimental): oral dexamethasone of 0.5mg/kg/day (max of 8mg/day), administered on post-operative days 1,3,5,7 in addition to standardized course of analgesics (opioids/acetaminophen/NSAIDs).
  Interventions: Drug: Dexamethasone; Drug: Analgesics
- analgesics alone (Active Comparator): standardized course of analgesics (opioids/acetaminophen/NSAIDs)
  Interventions: Drug: Analgesics

INTERVENTIONS:
Drug: Dexamethasone — dexamethasone solution or tablet (depending on age of patient) at 0.5mg/kg/day max of 8mg/day, administered on post-operative days 1,3,5,7.
  Arms: Dexamethasone plus analgesics
Drug: Analgesics — standardization of post-operative analgesics (narcotics and non-narcotic medication).
  * Oxycodone solution or tablet (depending on age of patient) at 0.05-0.1 mg/kg/dose every 6hrs; max 5mg (obese/OSA); prescribe 30 doses
  * Acetaminophen 10-15 mg/kg/dose every 6 hours; max 500mg per dose; prescribe 56 doses (over the counter medication)
  * Ibuprofen 5-10 mg/kg/dose every 6 hours; max 200 mg/dose; prescribe 56 doses (over the counter medication)

SUMMARY:
The purpose of this study is to determine if a post-operative course of oral dexamethasone affects opioid usage in pediatric patients undergoing tonsillectomy.

Patients who are scheduled to undergo tonsillectomy or adenotonsillectomy are randomized to receive either 1) a post-operative steroid course of oral dexamethasone in addition opioids, acetaminophen,NSAIDs or 2) opioids/acetaminophen/NSAIDS alone. All drugs are prescribed per approved FDA labeling. Children between the ages of 4-17 will be considered for enrollment.

Participants (or with the aid of parents/legal guardian for subjects unable to complete on their own) will complete a diary twice a day to record pain medication administration and visual pain scale. Remaining steroid and opioid medication will be measured at the routine post-operative appointment that occurs 4 - 6 weeks following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-17 years at time of surgery
* Scheduled for tonsillectomy or adenotonsillectomy surgery

Exclusion Criteria:

* Prior history of intracapsular tonsillectomy
* Previous diagnoses of Down Syndrome or developmental delay
* Presence of gastrostomy (g) tube
* A contraindication to steroids or steroid usage within 30 days prior to surgery including diabetes, allergy to steroid, already on chronic steroid, immune deficiency
* Active infection or concurrent operative procedures at the time of surgery
* Unable to read or speak English
* Pregnant or breastfeeding females

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2023-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Raynor, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center and affiliated practices, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexamethasone Plus Analgesics: oral dexamethasone of 0.5mg/kg/day (max of 8mg/day), administered on post-operative days 1,3,5,7 in addition to standardized course of analgesics (opioids/acetaminophen/NSAIDs).
  Dexamethasone: dexamethasone solution or tablet (depending on age of patient) at 0.5mg/kg/day max of 8mg/day, administered on post-operative days 1,3,5,7.
  Analgesics: standardization of post-operative analgesics (narcotics and non-narcotic medication).
  * Oxycodone solution or tablet (depending on age of patient) at 0.05-0.1 mg/kg/dose every 6hrs; max 5mg (obese/OSA); prescribe 30 doses
  * Acetaminophen 10-15 mg/kg/dose every 6 hours; max 500mg per dose; prescribe 56 doses (over the counter medication)
  * Ibuprofen 5-10 mg/kg/dose every 6 hours; max 200 mg/dose; prescribe 56 doses (over the counter medication)
- Analgesics Alone: standardized course of analgesics (opioids/acetaminophen/NSAIDs)
  Analgesics: standardization of post-operative analgesics (narcotics and non-narcotic medication).
  * Oxycodone solution or tablet (depending on age of patient) at 0.05-0.1 mg/kg/dose every 6hrs; max 5mg (obese/OSA); prescribe 30 doses
  * Acetaminophen 10-15 mg/kg/dose every 6 hours; max 500mg per dose; prescribe 56 doses (over the counter medication)
  * Ibuprofen 5-10 mg/kg/dose every 6 hours; max 200 mg/dose; prescribe 56 doses (over the counter medication)
Period: Overall Study
Arm/Group | Dexamethasone Plus Analgesics | Analgesics Alone
Started | 16 | 8
Completed | 14 | 7
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone Plus Analgesics | Analgesics Alone | Total
Number analyzed (Participants) | 16 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.8 (4.2) | 7.8 (2.7) | 8.5 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 8 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 7 | 19
  Unknown or Not Reported | 3 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 0 | 1 | 1
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Black or African American | 4 | 2 | 6
  Race: White | 12 | 4 | 16
  Race: More than one race | 0 | 0 | 0
  Race: Other | 0 | 1 | 1
  Race: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Opioid Use (Number of Doses)
Description: Measured by medication log and units remaining.
Time Frame: 4 weeks post-op
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Dexamethasone Plus Analgesics | Analgesics Alone
Number analyzed (Participants) | 14 | 7
doses | 11.5 (10.8) | 18.4 (8.4)
Statistical Analysis 1: Comparison: Dexamethasone Plus Analgesics vs Analgesics Alone; Test type: Equivalence — Test if the number of doses in Dexamethasone Plus Analgesics group differs from that in Analgesics Alone group at a significance level of 0.05; p = 0.16, t-test, 2 sided; Mean Difference (Final Values) = 6.9, 95% CI 2-sided [-2.9 to 16.7], Standard Deviation 10.1

2. Primary Outcome: Average Pain Score
Description: Measured by a visual analog scale, where 0 is no pain and 10 is worst possible pain.
Time Frame: 14 days post-op
Population: Participants who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexamethasone Plus Analgesics | Analgesics Alone
Number analyzed (Participants) | 14 | 7
score on a scale | 3.1 (1.7) | 2.7 (0.8)
Statistical Analysis 1: Comparison: Dexamethasone Plus Analgesics vs Analgesics Alone; Test type: Equivalence — Test if the average pain score in Dexamethasone Plus Analgesics group differs from that in Analgesics Alone group at a significance level of 0.05; p = 0.56, t-test, 2 sided; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.8 to 1.0], Standard Deviation 1.4

3. Secondary Outcome: Number of Participants With Post-operative Complications
Description: Post-op re-admissions and emergency room visits.
Time Frame: 30 days post-op
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone Plus Analgesics | Analgesics Alone
Number analyzed (Participants) | 14 | 7
Participants | 1 | 1
Statistical Analysis 1: Comparison: Dexamethasone Plus Analgesics vs Analgesics Alone; Test type: Equivalence — Test if the Number of participants with post-operative complications in Dexamethasone Plus Analgesics group differs from that in Analgesics Alone group at a significance level of 0.05; p = 1.00, Fisher Exact; Risk Difference (RD) = 0.07, 95% CI 2-sided [-0.22 to 0.36], Standard Error of Mean 0.15

ADVERSE EVENTS:
Time Frame: Up to 30 days post-op
Arm/Group | Dexamethasone Plus Analgesics | Analgesics Alone
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/8
Other Adverse Events (participants affected / at risk) | 12/16 | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone Plus Analgesics (N=16) | Analgesics Alone (N=8)
Emergency Room Visit (General disorders) | 1 | 1
Bleeding (Injury, poisoning and procedural complications) | 2 | 1
Nausea/Vomiting (Gastrointestinal disorders) | 5 | 3
Sleep Disturbance/Insomnia (General disorders) | 11 | 5
Fever (General disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Other - not specified (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT04541147/Prot_SAP_000.pdf